CLINICAL TRIAL: NCT00825422
Title: Assessment of Efficacy and Safety of Continuous Wound Infiltration With Local Anesthesics Through a Parietal Paravertebral Catheter for Postoperative Analgesia After Posterior Lumbar Arthrodesis
Brief Title: Local Anesthetic Infiltration to Prevent Postoperative Pain After Lumbar Surgery
Acronym: ICALP
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CHUBX 2008/21
Record Dates: First submitted 2009-01-19; First posted 2009-01-21 (Estimated); Last update posted 2012-06-20 (Estimated); Status verified 2012-06

CONDITIONS: Hyperalgesia
Keywords: Posterior lumbar arthrodesis; Degenerative spine; Postoperative analgesia; Local anesthesic; Continuous wound infusion catheter; Pain; lumbar vertebrae; Spinal fusion
MeSH Terms: conditions — Hyperalgesia; Pain | interventions — Ropivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): first bolus of 20 ml of ropivacaine(5mg/ml) and continuous infiltration (8ml/h)of ropivacaine (2mg/ml)
  Interventions: Drug: Ropivacaine / Placebo
- B (Placebo Comparator): first bolus of 20 ml of physiological saline solution(9%) and continuous infiltration (8ml/h)of physiological saline solution(9%)
  Interventions: Drug: Ropivacaine / Placebo

INTERVENTIONS:
Drug: Ropivacaine / Placebo — Wound infiltration with local anesthesics/placebo through a parietal paravertebral catheter

SUMMARY:
Posterior lumbar arthrodesis causes severe postoperative pain, hampering patients's postoperative reconvalescence especially functional rehabilitation. Efficient and safe methods for postoperative analgesia are, therefore, mandatory. The application of opioids are the most frequently used therapies for postoperative pain relief but it very often results side effects. Local anesthetic wound infiltration is widely recognized as a useful adjunct in a multimodal approach to postoperative pain management. In the setting of spine surgery, a single bolus administration of a local anesthetic is a useful method (with a reduction in parenteral morphine consumption during the 48 first hours) but has a limited effect because of its short duration of action. Prolonged administration through a multi-holed catheter positioned by the surgeon at the end of the procedure could increase the duration of action and may thereby improve the efficacy of local wound infiltration. Easy and effective, this new modality of administration has expanded the indications for parietal infiltrations toward major painful procedures.

We designed this study to determine whether local anesthetic (compared with saline solution) continuous wound infiltration during the first two days after posterior lumbar arthrodesis on degenerative spine, could improve postoperative analgesia at short-term but particularly at mid-term (two months) and long-term (six months), in order to decrease postoperative lumbar pains (resulting in best life quality, opioid consumption limited and rehabilitation hastened) and postoperative hyperalgesia areas. The postoperative analgesic and antihyperalgesic efficacies; the postoperative rehabilitation at mid-term and long term, and the safety of opioid administration and multi-holed parietal catheter will be compared in the two groups (control and study).

DETAILED DESCRIPTION:
Blockade of parietal nociceptive afferents by the use of continuous wound infiltration with local anesthetics may be beneficial in a multimodal approach to postoperative pain management after major surgery. The role of continuous wound parietal paravertebral infiltration of ropivacaine for pain relief and postoperative rehabilitation after posterior lumbar arthrodesis will be evaluated in a randomized, monocentric, double-blinded, superiority controlled trial.

The general purpose of this clinical research is the assessment of efficacy and safety of continuous wound infiltration with ropivacaine through a parietal paravertebral catheter for postoperative analgesia, and his repercussions at mid (two months) and long (six months)-term after posterior lumbar arthrodesis on degenerative spine.

The principal purpose concerns the assessment of postoperative analgesic efficacy at mid-term (two months after surgery) of continuous wound infiltration with ropivacaine (compared with saline solution), through a parietal paravertebral multi-holed catheter, after posterior lumbar arthrodesis.

After obtaining written informed consents, the patients scheduled to undergo posterior lumbar arthrodesis on degenerative spine,.will be randomly allocated to receive a continuous wound infusion of either 0.2% ropivacaine (ropivacaine group A) or 0.9% saline (control group B) when they will arrive in the operating room. The surgeon will perform a standardized posterior median incision at the level of lumbar intervertebral instability. Before putting retractors, he will infiltrate all surgical strata and the paraspinal muscles all long the wound bilaterally with a solution of ropivacaine 0.5% 20 mL (group A) or with a solution of 0,9% NaCl 20 ml (group B). At the end of surgery, a multi-holed wound catheter will be placed by the surgeon, under direct visualization, in the paravertebral space ; between the muscle fascia and subcutaneous tissues all along the wound, and fixed at the skin by a stitch. The patients will be thereafter randomly assigned to receive through the catheter either 0.2% ropivacaine (study group) (5-ml bolus followed by an infusion of 8 ml/h during 48 h) or the same protocol with 0.9% NaCl (control group), thanks to a prefilled elastomeric pump (400ml), set to deliver a 8-ml/h connected with the catheter. In addition, all patients will receive patient-controlled intravenous morphine analgesia. After the induction, the anaesthesist will install a peripheral venous catheter for each patient in order to make blood samples easier (eight peroperative and two postoperative blood samples for each patient, with the aim of ropivacaine pharmacokinetic study).

ELIGIBILITY:
Inclusion Criteria:

* Necessity to use safety contraceptive methods for women who can procreate
* Patients with American Society of Anesthesiologists physical status I, II or III
* Patients scheduled to undergo a posterior lumbar arthrodesis on one at three levels treated,
* Posterior lumbar arthrodesis is only executed on lumbar degenerative spine,
* A written informed consent has to sign by the patient and the investigator before beginning clinical study
* Patients affiliated with social security system

Exclusion Criteria:

* Pregnancy and breast-feeding
* Posterior lumbar arthrodesis exceeding three levels treated,
* Posterior lumbar arthrodesis post-traumatic or with neoplastic disorders or with the aim of correcting cord compression,
* Epilepsy not controlled through medication,
* Preoperative cognitive dysfunction or psychiatric disorders,
* Cardiac or breathing dysfunctions,
* Preoperative opioid consumption,
* Patients who have a known local anesthetic, or morphine or/and acetaminophen allergy,
* Lack of understanding about the study or inability to use the patient controlled analgesic device,
* Patients protected by the law, guardianship,
* Patients who take a share in an another clinical study in the same time,

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2009-01; Primary Completion 2010-04 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Postoperative pain score : Visual Analog Scale (VAS) | Two months after surgery

SECONDARY OUTCOMES:
Blood dosages of total ropivacaine | Peroperative
Clinical tolerances of catheter | until 5 days after surgery
Pain score :visual analog scale (VAS) | 24h, 48h, 5 days, 2 and 6 months after surgery
Static hyperalgesia using von Frey filaments | 48h, 5 days, 2 and 6 months after surgery
Postoperative rehabilitation neuropathic pain | 2 and 6 months after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Geneviève CHENE, Professor, Study Chair — University Hospital, Bordeaux; Cécile DEGRYSE, MD, Principal Investigator — Univestity Hospital, Bordeaux
Locations (1):
- University Hospital, Bordeaux, France